CLINICAL TRIAL: NCT02808273
Title: Use of Bemiparine as a Prophylactic Antitrombotic Agent, in Patients Undergoing Microsurgery for Head and Neck Reconstruction
Brief Title: Use of Bemiparine as a Prophylactic Antithrombotic Agent, in Patients Undergoing Microsurgery for Head and Neck Reconstruction
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: FUN-BEM-2015-01
Record Dates: First submitted 2016-03-04; First posted 2016-06-21 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2018-02

CONDITIONS: Patients Undergoing Microvascular Surgery
Keywords: Bemiparine; Antithrombotic microsurgery protocol; Comparative study; Anticoagulant microsurgery protocol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective control: Patients who had received enoxaparine as antithrombotic according to a protocol for prevention of postoperative deep venous thrombosis
- Prospective Cohort: Patients who will receive bemiparine 3500 UI as antithrombotic according to a protocol for prevention of postoperative deep venous thrombosis
  Interventions: Drug: Bemiparine

INTERVENTIONS:
Drug: Bemiparine — Bemiparine 3500 UI as antithrombotic according to a protocol for prevention of postoperative deep venous thrombosis
  Other Names: Hibor (3500UI/0,2ml)
  Groups: Prospective Cohort

SUMMARY:
A comparative study to reveal if the use of Bemiparine (Hibor) versus Enoxaparin (Clexane) as an antithrombotic agent, shows an advantage on the rate of thrombotic and haemorrhagic events in microsurgicals free flaps during head and neck reconstruction.

DETAILED DESCRIPTION:
This is an observational post-authorization study on a group of patients undergoing microsurgery on the Oral and Maxillofacial Surgery and Plastic and Reconstructive Surgery Service at Ramon y Cajal Hospital, Madrid for processes that require reconstruction with a flap microvascular. A group of 67 patients treated according protocol postoperative prevention of deep vein thrombosis with Bemiparina will be compared with data collected retrospectively from a group of 134 patients treated previously with an earlier protocol with enoxaparin as main antithrombotic agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will undergo reconstructive surgery for defects in any part of the body, especially in head and neck, after cancer, traumatic or infectious pathology, which will require the use of techniques of microsurgery.
* Patients who have given their informed consent
* Patients in which it has been decided to use thromboprophylaxis with bemiparina before proposing them to participate in the study.

Exclusion Criteria:

* Patients not eligible for repair through the use of free flaps, and therefore the use of Microsurgical techniques for vascular anastomosis
* Patients with an underlying pathology that may interfere to a clinically significant or contraindicated the use of Bemiparina, such as: serious hepatic or renal insufficiency, uncontrolled arterial hypertension, history of gastroduodenal, thrombocytopenia, nephrolithiasis or uretrolitiasis and vascular disease ulcer of choroid and retina.
* Refusal of the patient or their family members to participate in the study.
* Pregnancy and breastfeeding
* Known hypersensitivity to study drugs or any of its components

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who will undergo Oral and Maxillofacial or Plastic surgery that require reconstruction with microvascular flap at Hospital Ramón y Cajal, Madrid. A group of 67 patients treated according to a protocol for prevention of postoperative deep venous thrombosis with Bemiparina that will be compared with data collected from a group of 134 patients previously treated with a similar protocol but enoxaparin as antithrombotic agent.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
To compare the use of Bemiparine, against Clexane as an antithrombotic agent | 24 months
  Incidence thrombotic complications and bleeding

SECONDARY OUTCOMES:
Incidence of deep vein thrombosis and pulmonary embolism | 24 months
Incidence of postsurgery hemorrhagic strokes with both drugs | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Julio Acero Sanz, MD; PhD, Principal Investigator — Ramon y Cajal Hospital
Locations (1):
- Ramon y Cajal Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No